CLINICAL TRIAL: NCT01428570
Title: Comparison of the Pentax AWS® With the Macintosh Laryngoscope for Tracheal Intubation in Patients With Obstructive Sleep Apnea Syndrome: a Randomized Comparative Study
Brief Title: Comparison of the Pentax AWS® With the Macintosh Laryngoscopic Intubation in Obstructive Sleep Apnea Syndrome Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Mi Kyeong Kim, Assistant Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PEN
Record Dates: First submitted 2011-08-31; First posted 2011-09-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Sleep Apnea, Obstructive
Keywords: sleep apnea, obstructive; intubation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentax-AWS (Experimental): Patients in this group will be intubated using Pentax-AWS
  Interventions: Device: Pentax-AWS (AWS; Pentax Corporation, Tokyo, Japan)
- laryngoscopy (Active Comparator): Patients in this group will be intubated using Macintosh laryngoscope.
  Interventions: Device: Pentax-AWS (AWS; Pentax Corporation, Tokyo, Japan)

INTERVENTIONS:
Device: Pentax-AWS (AWS; Pentax Corporation, Tokyo, Japan) — Each group of patients will be intubated using the Macintosh laryngoscope or Pentax-AWS.

SUMMARY:
The Pentax-AWS_ system (AWS; Pentax Corporation, Tokyo, Japan) is a new rigid indirect laryngoscope which has an integrated tube passage function. Pentax-AWS improved the laryngeal view and facilitated tracheal intubation in patients with restricted neck motion. The purpose of this clinical trial was to evaluate the relative efficacy of the AWS laryngoscopes when used by experienced anesthetists in Obstructive Sleep Apnea Syndrome (OSAS) patients and to compare its performance with the Macintosh laryngoscope.

DETAILED DESCRIPTION:
The occurrence of difficult intubation in OSAS patients is higher than in age and sex matched control patients. The Pentax-AWS_ system (AWS; Pentax Corporation, Tokyo, Japan) is a new rigid indirect laryngoscope which has an integrated tube passage function. Several studies reported that Pentax-AWS improved the laryngeal view and guide also facilitated rapid, easy and reliable tracheal intubation in patients undergoing elective surgery. The purpose of this clinical trial was to evaluate the relative efficacy of the AWS laryngoscopes when used by experienced anesthetists in OSAS patients and to compare its performance with the Macintosh laryngoscope. The investigators hypothesized that, in comparison with the Macintosh, AWS would reduce intubation difficulty, as measured by the intubation difficulty scale (IDS) score.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3 patients,
* aged 20years or older,
* undergoing uvulopalatopharyngoplasty(UPPP) surgery under general anesthesia for a polysomnography-confirmed diagnosis of OSAS.

Exclusion Criteria:

* unstable teeth or mouth opening of < 18mm
* Patients with any pathology of the neck,
* upper respiratory tract or upper alimentary tracts,
* risk of pulmonary aspiration of gastric contents,
* a history of relevant drug allergy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Intubation Difficulty Scale(IDS) score | After the end of intubation (within 10 minute after the end of intubation.)
  IDS score will be recorded within 10 minute after the end of intubation.

SECONDARY OUTCOMES:
Cormack and Lehane grade | After the end of intubation (within 10 minute after the end of intubation.)
  Cormack and Lehane grade will be recorded within 10 minute after the end of intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Mi Kyeong Kim, Professor, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee university hospital, Seoul, South Korea